CLINICAL TRIAL: NCT06496828
Title: Clinical Performance of All-Ceramic Crowns on Teeth Prepared With Biologically Oriented Preparation Technique Compared to Horizontal Preparation
Brief Title: Clinical Outcomes of Biologically Oriented Preparation Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Prosthodontics-01-2024
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Crowns; Tooth Preparation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biologically-oriented preparation technique (BOPT) (Experimental): Patients in this group will undergo the biologically-oriented preparation technique.
  Interventions: Procedure: Biologically-oriented preparation technique
- Conventional preparation (Active Comparator): Patients in this group will undergo the convention preparation technique.
  Interventions: Procedure: Conventional method of preparation

INTERVENTIONS:
Procedure: Biologically-oriented preparation technique — The preparation will be made according to the new principles of biologically oriented technique to receive monolithic and bi-layered all-ceramic crowns.
  Arms: Biologically-oriented preparation technique (BOPT)
Procedure: Conventional method of preparation — Teeth prepared with shoulder margins to receive monolithic and bi-layered all-ceramic crowns
  Arms: Conventional preparation

SUMMARY:
This study aims to evaluate the periodontal response of teeth prepared with a biologically oriented preparation technique (BOPT) compared to conventional preparation for all-ceramic crowns.

DETAILED DESCRIPTION:
The study aims to evaluate the clinical performance of all-ceramic crowns on teeth prepared with two different types of preparations.

This randomized controlled trial will include 60 teeth divided into two groups: 30 teeth will be prepared with BOPT, and 30 teeth will be prepared with shoulder margins. All teeth will receive monolithic or bi-layered ceramic crowns.

Patients are planned to attend follow-up visits after 3, 6, 12, and 18 months, respectively, after cementation. Probing depth, gingival recession, bleeding on probing, gingival index, gingival thickness, patient opinion, and mechanical and biological complications are all recorded at check-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18.
* Two teeth at least needed to be restored with full crowns (each patient needs at least two single crowns).
* Stable occlusion.
* Good oral hygiene.
* Periodontally healthy teeth.
* Nonsmoking or smoking less than ten cigarettes/day.
* Probing depth between 1 and 3 mm.

Exclusion Criteria:

* Patients younger than 18.
* Parafunctional habits.
* Active periodontal disease.
* Poor oral hygiene.
* Systemic disease that may affect the periodontal health.
* Pregnancy.
* Radiation or chemotherapy.
* Treatment by Bisphosphonates medication.
* Patients who are unable or unwilling to attend follow-up visits

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Plaque index | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation of the crowns.
  The plaque index will be measured at the buccal, lingual, mesial, and distal sites of each included tooth, according to Löe and Silness, 1963
Change in the gingival index | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation of the crowns.
  The gingival index will be measured at the buccal, lingual, mesial, and distal sites of each included tooth according to Silness and Löe, 1964
Change in the probing depth | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation of the crowns.
  A UNC periodontal probe will be used to measure the probing depth at the buccal, lingual, mesial, and distal sites of each included tooth.
Change in bleeding on probing | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation of the crowns.
  This variable will be measured at the buccal, lingual, mesial, and distal sites of each included tooth, recorded simultaneously with probing depth, according to Ainamo and Bay, 1975
Change in the gingival marginal stability | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation of the crowns.
  The gingival marginal stability at the buccal site will be measured using a UNC periodontal probe and a transparent jig to measure the distance between a reference point on the jig and the free gingival margin.
Change in the free gingiva thickness | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation of the crowns.
  The free gingiva thickness will be measured at the buccal site using a transparent jig with a reference point on the marginal gingiva, a 15-size spreader with a rubber stopper, and a millimetric ruler

SECONDARY OUTCOMES:
Change in the internal and marginal adaptation | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation.
  The internal and marginal adaptation will be dong using the replica technique. It will be carried out after clinical assessment and cementation of all crowns. An in vitro study utilizing an optical microscope with a micron-graded ruler will be implemented.
Change in the functional and mechanical complications | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation.
  The functional and mechanical complications will be appraised. The existence of cracks, chipping, and/ or fracture of crowns and their size if exist according to FDI criteria (Hickel et al., 2010) will be evaluated.
Change in the secondary caries status | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation.
  The secondary caries status will be assessed according to Cvar and Ryge, 2005. The presence or absence of caries at the cervical margins of the abutments will be recorded. Other biological complications, such as abutment fracture, root fracture, and/ or pulpitis will be reported, too
Change in the marginal adaptation after crown cementation | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation.
  The marginal adaptation after crown cementation will be clinically evaluated using a sharp dental probe, according to Cvar and Ryge, 2005, at each follow-up appointment.
Change in the color matching | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation.
  The level of color matching will be assessed according to Cvar and Ryge (2005). To measure this outcome, color matching with adjacent teeth, slight mismatching, or major mismatching of color and/or translucency will be reported.
Change in the clinical success | Will be recorded at 1 week, 1, 3, 6, 12, and 18 months after cementation.
  The clinical success status will be assessed according to Walton, 2002. This outcome will be evaluated in case any patient cannot attend the follow-up visits during the trial for any reason. Thus, success might be evaluated indirectly by a phone call if possible.
Change in patients' satisfaction | This will be measured at one week and 18 months following cementation.
  Patients' satisfaction will be assessed according to FDI criteria (Hickel et al., 2010). This outcome will report the level of patient satisfaction functionally and aesthetically. Complete satisfaction, light criticism, major criticism, and entirely dissatisfaction are the levels of the patient's view that will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Aljareh, DDS MSc, Principal Investigator — Department of Fixed Prosthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria; Nabil Alhouri, DDS MSc PhD, Study Director — Department of Fixed Prosthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria; Mohanad Kadhim, DDS MSc PhD, Study Director — Department of Periodontology, Faculty of Dentistry, Iraq.
Locations (1):
- Department of Fixed Prosthodontics, University of Damascus Dental School, Damascus, Syria, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohammad A, Abraham S, Nada A. The effect of biologically oriented and subgingival horizontal preparation techniques on periodontal health: A double-blind randomized controlled clinical trial. Saudi Dent J. 2023 Sep;35(6):727-733. doi: 10.1016/j.sdentj.2023.06.003. Epub 2023 Jun 17. PMID 37817795
- [Background] Palombo D, Rahmati M, Vignoletti F, Sanz-Esporrin J, Salido MP, Haugen HJ, Sanz M. Hard and soft tissue healing around teeth prepared with the biologically oriented preparation technique and restored with provisional crowns: An in vivo experimental investigation. J Clin Periodontol. 2023 Sep;50(9):1217-1238. doi: 10.1111/jcpe.13825. Epub 2023 May 30. PMID 37253614
- [Background] Agustin-Panadero R, Serra-Pastor B, Loi I, Suarez MJ, Pelaez J, Sola-Ruiz F. Clinical behavior of posterior fixed partial dentures with a biologically oriented preparation technique: A 5-year randomized controlled clinical trial. J Prosthet Dent. 2021 Jun;125(6):870-876. doi: 10.1016/j.prosdent.2020.03.031. Epub 2020 Jun 21. PMID 32580920
- [Background] Serra-Pastor B, Bustamante-Hernandez N, Fons-Font A, Fernanda Sola-Ruiz M, Revilla-Leon M, Agustin-Panadero R. Periodontal Behavior and Patient Satisfaction of Anterior Teeth Restored with Single Zirconia Crowns Using a Biologically Oriented Preparation Technique: A 6-Year Prospective Clinical Study. J Clin Med. 2021 Aug 6;10(16):3482. doi: 10.3390/jcm10163482. PMID 34441778
- [Background] Agustin-Panadero R, Serra-Pastor B, Fons-Font A, Sola-Ruiz MF. Prospective Clinical Study of Zirconia Full-coverage Restorations on Teeth Prepared With Biologically Oriented Preparation Technique on Gingival Health: Results After Two-year Follow-up. Oper Dent. 2018 Sep/Oct;43(5):482-487. doi: 10.2341/17-124-C. Epub 2018 Mar 7. PMID 29513640
- [Background] Paniz G, Nart J, Gobbato L, Chierico A, Lops D, Michalakis K. Periodontal response to two different subgingival restorative margin designs: a 12-month randomized clinical trial. Clin Oral Investig. 2016 Jul;20(6):1243-52. doi: 10.1007/s00784-015-1616-z. Epub 2015 Oct 8. PMID 26445857
- [Background] Loi I, Di Felice A. Biologically oriented preparation technique (BOPT): a new approach for prosthetic restoration of periodontically healthy teeth. Eur J Esthet Dent. 2013 Spring;8(1):10-23. PMID 23390618